CLINICAL TRIAL: NCT02065843
Title: Comparative Study of the Effectiveness of Three Anxiolytic Drugs Used in Third Molar Surgery
Brief Title: Three Anxiolytic Drugs Used in Third Molar Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal de Sergipe (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Liane Maciel de Almeida Souza, Professor, Universidade Federal de Sergipe
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANSI-388.427
Record Dates: First submitted 2014-02-15; First posted 2014-02-19 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Dental Anxiety; Impacted Third Molar Tooth
Keywords: Anxiety; Third molar surgery; Blood pressure; Heart rate; Oxygen saturation
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mulungu (Active Comparator): 500 mg Mulungu Matusa® (Erytrina mulungu, 2 capsules of 250 mg) to be administered v.o., one hour before the surgical procedure.
  Interventions: Drug: Mulungu
- placebo (Placebo Comparator): 500 mg of starch (2 capsules of 250 mg) to be administered v.o., one hour before the surgical procedure.
  Interventions: Drug: Placebo
- Passiflora incarnata (Active Comparator): 100 mg Passiflora incarnata (2 capsules of 50 mg) to be administered v.o., one hour before the surgical procedure.
  Interventions: Drug: Passiflora incarnata
- midazolam (Active Comparator): 15 mg midazolam (2 capsules of 7.5 mg) to be administered v.o., one hour before the surgical procedure.
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: Mulungu — 500 mg/single dose/1 hour before dental surgery
  Other Names: Mulungu Matusa, Erytrina mulungu
  Arms: Mulungu
Drug: Placebo — 500 mg/single dose/1 hour before dental surgery
  Arms: placebo
Drug: Passiflora incarnata — 100 mg/single dose/1 hour before dental surgery
  Arms: Passiflora incarnata
Drug: midazolam — 15 mg/single dose/1 hour before dental surgery
  Other Names: Dormonid
  Arms: midazolam

SUMMARY:
This study was to compare the effectiveness of three drugs (Passiflora incarnata, Erythrina mulungum, Midazolam) in controlling anxiety in patients undergoing bilateral extraction of asymptomatic, impacted mandibular third molars.

DETAILED DESCRIPTION:
In this research, characterized as a randomized, double-blind, parallel study, 200 healthy volunteered patients aging 18 or older will be distributed into 4 groups (n=50) as follows: Group I - 500mg Erythrina mulungu; Group II - placebo; Group III ; 100 mg Passiflora incarnata; Group IV - 15 mg midazolam. All treatments will be administered p.o. 1 hour randomly prior to the surgical procedures. The level of anxiety will be assessed through questionnaires and physical parameters, such as blood pressure, heart rate and oxygen concentration in three periods: at baseline, right before the surgical procedures and after 7 days. Data will be collected, tabulated and analyzed by the following statistical tests: chi-square, t-test, ANOVA and Tukey test, Friedman, Fisher's exact test with significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* indication of bilateral extraction of asymptomatic, impacted mandibular third molars

Exclusion Criteria:

* patients under the age of 18 any general health problem based on the medical history and physical examination history of use of any medication within 15 days before the beginning of the research history of hypersensitivity to drugs, substances or materials used in this experiment pregnancy or lactation history of pericoronitis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in anxiety report | Change from baseline to 7 days
  Changes in the subjects' anxiety level will be observed by using a Modified Corah Dental Anxiety Scale in three times: at baseline, in the day of surgery and after 7 days of the procedure.

SECONDARY OUTCOMES:
Changes in blood pressure | Change from baseline to 2 hours
  blood pressure (mmHg) will be measured before the drugs administration, 30 minutes after drugs administration and during local anesthesia, incision, tooth removal and suturing.
Changes in heart rate | Change from baseline to 2 hours
  heart rate (bpm) will be measured before drugs administration, 30 minutes after drugs administration and during local anesthesia, incision, tooth removal and suturing.
Changes in oxygen saturation | Change from baseline to 2 hours
  oxygen saturation (SpO2) will be measured before drugs administration, 30 minutes after drugs administration and during local anesthesia, incision, tooth removal and suturing.

CONTACTS AND LOCATIONS:
Overall Officials: Liane M Souza, PhD, Principal Investigator — Federal University of Sergipe
Locations (1):
- Federal University of Sergipe, Aracaju, Sergipe, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will be kept not available

REFERENCES:
- [Background] Balbani AP, Silva DH, Montovani JC. Patents of drugs extracted from Brazilian medicinal plants. Expert Opin Ther Pat. 2009 Apr;19(4):461-73. doi: 10.1517/13543770902824180. PMID 19441926
- [Background] Flausino OA Jr, Pereira AM, da Silva Bolzani V, Nunes-de-Souza RL. Effects of erythrinian alkaloids isolated from Erythrina mulungu (Papilionaceae) in mice submitted to animal models of anxiety. Biol Pharm Bull. 2007 Feb;30(2):375-8. doi: 10.1248/bpb.30.375. PMID 17268084
- See also: published article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4192578/pdf/medoral-19-e518.pdf